CLINICAL TRIAL: NCT04188574
Title: A Multi-Centre, International, Randomised, Vehicle Controlled, Parallel-Group, Double-Blinded Phase 2 Trial of BB2603 Topical Treatment in Subjects With Distal Subungual Onychomycosis (DSO) of the Toenail
Brief Title: A Trial Involving Treatment of BB2603 in Subjects With Distal Subungual Onychomycosis of the Toenail
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Blueberry Therapeutics (Industry)
Collaborators: IQVIA Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BBTAF202
Record Dates: First submitted 2019-09-16; First posted 2019-12-06 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Distal Subungual Onychomycosis; Fungal Infection; Fungus, Nail
Keywords: DSO; Fungual Infection; Fungus, Nail
MeSH Terms: conditions — Mycoses; Onychomycosis

STUDY DESIGN:
Intervention Model Description: Double-Blinded
Who Masked: Participant, Investigator
Masking Description: Treatment allocation will not be disclosed to the site team or subject or the clinical Sponsor team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BB2603-10 (Experimental): Treatment with topical spray twice-daily (BID) BB2603-10: 0.1% terbinafine
  Interventions: Drug: BB2603-10; Other: Vehicle
- BB2603-3 (Experimental): Treatment with topical spray twice-daily (BID) BB2603-3: 0.03% terbinafine
  Interventions: Drug: BB2603-3; Other: Vehicle
- BB2603-1 (Experimental): Treatment with topical spray twice-daily (BID)BB2603-1: 0.01% terbinafine
  Interventions: Drug: BB2603-1; Other: Vehicle
- Vehicle Control (Other): 0.3% polyhexanide/ 20% ethanol/ water formulation.
  Interventions: Drug: BB2603-1; Drug: BB2603-3; Drug: BB2603-10; Other: Vehicle

INTERVENTIONS:
Drug: BB2603-1 — Treatment with topical spray twice-daily (BID) BB2603-1: 0.01% terbinafine
  Arms: BB2603-1; Vehicle Control
Drug: BB2603-3 — Treatment with topical spray twice-daily (BID) BB2603-3: 0.03% terbinafine
  Arms: BB2603-3; Vehicle Control
Drug: BB2603-10 — Treatment with topical spray twice-daily (BID) BB2603-10: 0.1% terbinafine
  Arms: BB2603-10; Vehicle Control
Other: Vehicle — Treatment with topical spray twice-daily (BID): 0.3% polyhexanide/ 20% ethanol/ water formulation.

SUMMARY:
This study will be a multicenter, international, randomized, vehicle-controlled, parallel-group, double-blinded study. Subjects who are eligible to participate with a confirmed diagnosis of Distal Subungual onychomycosis (DSO) of the toenail will be randomized and participate in one of the following treatment groups: BB2603-1: 0.01% terbinafine/0.03% polyhexanide formulation, or BB2603-3: 0.03% terbinafine/0.09% polyhexanide formulation, or BB2603-10: 0.1% terbinafine/0.3% polyhexanide formulation, or Vehicle: 0.3% polyhexanide/20% ethanol/water formulation. The subject in each treatment group will be treated twice daily (BID) for 12 weeks and then complete a 28-day post-treatment visit.

DETAILED DESCRIPTION:
Onychomycosis (OM; fungal nail infection) is a common and contagious fungal infection of the nail plate or nail bed, leading to the gradual destruction of the nail plate. OM is considered the most prevalent of the nail ailments, accounting for about 50% of all diseased nails and about 30% of cutaneous fungal infections. The prevalence of OM is reported to be 23% across Europe, 13.8% in North America and approximately 10% in Japan, with the prevalence increasing in Western countries, presumably due to lifestyle changes and the ageing of the population.

Distal subungual onychomycosis (DSO) is the most common form of OM, characterised by invasion of the nail bed and underside of the nail plate beginning at the hyponychium. This infection is visualised as nails with normal surface texture and thickness but variable "bays" of white nail that extend from the distal nail tip proximally into the area of the nail bed. The vast majority of cases of OM are caused by dermatophyte fungi. In 80% to 98% of affected individuals, Trichophyton rubrum with additional infections caused by Trichophyton mentagrophytes var interdigitale (commonly referred to as Trichophyton mentagrophytes) or Epidermophyton floccosum. The dermatophyte Trichophyton rubrum is the major cause of tinea pedis (TP; athlete's foot) and OM. OM is a progressive disease; if left untreated, OM can lead to permanent nail damage and associated discomfort.

Onychomycosis is currently treated with surgery, medical devices (eg laser therapy), oral or topical anti-fungal agents or a combination of both. Oral terbinafine, when used for a minimum of 3 months, can achieve an efficacy of 38% or higher if treatment is extended but has a significant drug-interaction and side effect profile, including liver failure, and periodic monitoring (after 4-6 weeks of treatment) of liver function test is recommended. Topical agents are used for up to 18 months but have significantly lower efficacy rates of less than 20%.

Terbinafine is a well-established synthetic allylamine anti-fungal developed by Sandoz (now Novartis) and commercially available worldwide for more than 25 years in different oral and topical formulations as a dermal cream (1%), emulsion gel (1%), solution/spray (1%), as well as oral tablets (250 mg and 125 mg). It is highly hydrophobic in nature and tends to accumulate in skin, nails, and fatty tissues. Terbinafine's anti-fungal mechanism of action is by inhibition of squalene epoxidase in the fungal cell membrane. This leads to a deficiency in ergosterol and an intracellular accumulation of squalene, resulting in fungal cell rupture/lysis (fungicidal activity).

Dermatophytoses of nails, in contrast to those at other body sites, are particularly difficult to eradicate with drug treatment. This is the consequence of factors intrinsic to the nail (the hard, protective nail plate, sequestration of pathogens between the nail bed and plate, and slow growth of the nail). The unique barrier properties of the nail plate, which hampers the passage of anti-fungal drugs in a concentration required to eradicate the deeply-seated causative fungi in the nail bed, is a specific challenge.

As such, there is a recognized need for a simple, effective and curative topical treatment for OM. Furthermore, topical treatment may result in minimal adverse systemic events and possibly improved adherence.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 (and ≤99) at the time of Informed Consent.
2. Clinically and mycologically (KOH and culture positive for dermatophytes [microbial infection with fungus belonging to the genus Trichophyton, Microsporum, Epidermophyton]) confirmed diagnoses of DSO of the target toenail affecting ≥25% to ≤60% of the target toenail as determined through clinimetric measurement.
3. Signed written informed consent form (ICF) prior to any trial related activity (subjects must have the mental, literate, and legal ability to give a written informed consent, which must comply with the ICH GCP guidelines and local requirements).
4. Subjects must be willing and able to comply with trial requirements.
5. Females must be either postmenopausal for ≥1 year (ie 12 consecutive months of amenorrhea, for which there is no other obvious pathologic or physiologic cause), or surgically sterile (tubal ligation, hysterectomy, or bilateral oophorectomy) for at least 6 months or, if of childbearing potential must use either highly effective birth control methods such as:

   * Oral, intravaginal or transdermal oestrogen- and progestogen-containing hormonal contraception associated with inhibition of ovulation
   * Oral, injectable or implantable progestogen-only hormonal contraception associated with inhibition of ovulation
   * Intrauterine device or intrauterine hormone-releasing system
   * Bilateral tubal occlusion
   * Vasectomised partner provided that the partner is the sole sexual partner and that the vasectomised partner has received medical assessment of the surgical success Clinical Study Protocol
   * Sexual abstinence, ie, refraining from heterosexual intercourse during the entire period of risk associated with the trial treatments

OR

Acceptable birth control methods such as:

* Progestogen-only oral hormonal contraception, where inhibition of ovulation is not the primary mode of action
* Male or female condom with or without spermicide
* Cap, diaphragm or sponge with spermicide
* A combination of male condom with either cap, diaphragm or sponge with spermicide (double barrier methods) are also considered acceptable birth control methods

while using trial medication and 28 days after last dose of IMP.

Birth control methods which are considered unacceptable: Periodic abstinence (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhoea method. Female condom and male condom should not be used together.

Treatment with the IMP will be discontinued in case of pregnancy.

The criteria with respect to pregnancy and contraception are in line with the CTFG Recommendations, v1.1, Sept 2020.

Exclusion Criteria:

1. Any other form of OM except DSO.
2. Nails with clinical evidence of no or low distal growth.
3. DSO of the target toenail where involvement has extended into the proximal portion of the target nail (unaffected proximal nail is ≤3mm) or nail matrix. Any severe OM defined as 3 or more affected toes on one foot.
4. Estimated target toenail thickness >3mm.
5. Presence of dermatophytoma (defined as thick masses of fungal hyphae and necrotic keratin between the nail plate and nail bed) on the target nail.
6. History of dermatophyte infections unresponsive to systemic or topical anti-fungal drugs (other than OM).
7. Presence of toenail infection that does not involve a dermatophyte.
8. Presence of toenail infection that involves a non-dermatophyte fungus or yeast in combination with a dermatophyte, where the non-dermatophyte is, in the opinion of the Investigator, considered to be causative of OM based on clinical appearance, medical history or lifestyle risk.
9. Topical treatment with an antifungal medication within 12 weeks before Randomisation/Visit 2 (with the exception of up to 2 weeks' treatment during the screening period with a non-terbinafine topical antifungal to treat clinically active TP).

   Other exclusion criteria
10. Systemic use of anti-fungal treatment within 12 months before Randomisation/Visit 2.
11. Past use within the last 6 months before Randomisation/Visit 2 or planned use of laser therapy, photodynamic therapy, chemical, surgical, relevant mechanical removal for OM or debridement.
12. Concomitant clinically suspected active TP at Randomisation/Visit 2.
13. Known allergy or known intolerabilities to any of the tested treatment products.
14. Subjects with diabetes, immune suppression, peripheral vascular disease, lymphatic insufficiency, recurrent cellulitis, or other compromised states of health whether due to underlying medical disorders or to long-term immunosuppressive treatments (including >4 weeks systemic corticoids or >4 weeks topical corticoids on the feet). Topical immunosuppressive treatment if not on the target nail is allowed.
15. Females of childbearing potential with a positive serum pregnancy test at Screening/Visit 1 and/or a positive urine pregnancy test at Randomisation/Visit 2 are excluded.
16. Women of childbearing potential who are pregnant or breast feeding or who plan to become pregnant after enrolment until 28 days after the last dose of IMP.
17. Subjects previously randomised in this trial or received BB2603 previously.
18. Use of any investigational agent during the study or within 28 days or 5 half-lives prior to Randomisation/Visit 2, whichever is longer.
19. Close affiliation with the Investigator (eg, a close relative) or persons working at a trial site, or subject who is an employee of the Sponsor's company.
20. Subjects who are institutionalised because of legal or regulatory order.
21. Hepatic impairment with AST or ALT >5 x Upper Limit of Normal.
22. Estimated creatinine clearance using Cockcroft-Gault formula and actual body weight <30 ml/min.
23. Presence of any other condition or infection of the foot or nail or other disease process that might affect the safety and well-being of the subject or confound the treatment evaluation (eg, psoriasis, lichen planus, or other medical conditions known to induce nail changes, trauma, previous toenail surgery with any residual disfigurement or any dermatological or nail condition that could mimic the signs and symptoms of OM, signs of severe peripheral circulatory insufficiency, use of chronic immunosuppressive medication or radiation therapy within 2 months prior to trial entry or planned during the trial period, immunocompromised).
24. Subjects deemed to be at risk of re-infection or recurrence of OM due to occupational, environmental or behavioural lifestyle in the opinion of the Investigator.
25. Any other significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in this trial, or may influence the result of the trial, or the subject's availability to participate in the trial.
26. Any known or suspected hypersensitivity to, or known allergy to, or other intolerability to BB2603 or its active ingredient or excipients.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Number of subjects with an Early Response for BB2603-10 versus vehicle | 16 weeks
  Early Response is defined as clinimetrically assessed clear nail growth (yes/no) and/or negative dermatophyte culture (yes/no).

SECONDARY OUTCOMES:
Number of subjects with a Complete Cure for BB2603-10 versus vehicle | 52 weeks
  Complete Cure is assessed programmatically and is defined as satisfying the following: binary (yes/no) completely clear nail and mycological response (negative KOH and negative dermatophyte culture).
Number of subjects with Completely Clear Nail, Almost Clear Nail, Negative KOH or Negative Dermatocyte Culture, assessed separately, for BB2603-10 versus vehicle | 52 weeks
  Completely Clear Nail (yes/no), Almost Clear Nail (yes/no), Negative KOH (yes/no) and Negative Dermatocyte Culture (yes/no) are each assessed separately
Concentration of terbinafine in the plasma in all subjects | 52 weeks
  Terbinafine, the active component of BB2603, will be measured in pg/ml
Number of subjects with adverse events | 16, 24, 28 weeks
  Safety and tolerability data will be assessed by number of subjects with adverse events (AEs), serious adverse events, drug discontinuations due to AEs, and deaths. Data will be assessed at Week 16, 24 and 28 .
Number of subjects with an Early Response for BB2603-1 or BB2603-3, respectively versus vehicle | 16 weeks
  Early Response is defined as clinimetrically assessed clear nail growth (yes/no) and/or negative dermatophyte culture (yes/no).
Number of subjects with a Complete Cure for BB2603-1 or BB2603-3, respectively versus vehicle | 52 weeks
  Complete Cure is assessed programmatically and is defined as satisfying the following: binary (yes/no) completely clear nail and mycological response (negative KOH and negative dermatophyte culture).
Number of subjects with Completely Clear Nail, Almost Clear Nail, Negative Dermatocyte Culture or Negative Dermatophyte Culture, assessed separately for BB2603-1 or BB2603-3, respectively versus vehicle | 52 weeks
  Completely Clear Nail (yes/no), Almost Clear Nail (yes/no), Negative KOH (yes/no) and Negative Dermatocyte Culture (yes/no) are each assessed separately

CONTACTS AND LOCATIONS:
Locations (20):
- Czechia (2):
  - Dermatovenerologická klinika VFN, Prague
  - Sanatorium prof. Arenbergera, Prague
- Germany (6):
  - Licca Clinical Research Institute, Augsburg
  - Praxis Dr. med. Thomas Wildfeuer & Kolleg*innen, Berlin
  - Hautzentrum Jahrhunderthaus Gemeinschaftspraxis Dres. Niesmann und Othlinghaus, Bochum
  - Uniklink Carl Gustav Carus, Klinik und Polyklinik für Dermatologie, Dresden
  - Hautarztpraxis Dres. Leitz, Stuttgart
  - Centroderm GmbH, Wuppertal
- Poland (12):
  - NZOZ Dermal, Bialystok
  - NZOZ Osteo-Medic, Bialystok
  - Klinika Dermatologii, Wenerologii, Gdansk
  - Centrum Medyczne Angelius Provita, Katowice
  - Gyncentrum Osrodek Badan Klinicznych, Katowice
  - ETG Lodz, Lodz
  - Etg Lublin Kunickiego, Lublin
  - ETG Siedlce, Siedlce
  - Laser Clinic, Szczecin
  - ETG Warszawa, Warsaw
  - dermMedica, Wroclaw
  - ETG Zamość, Zamość

IPD SHARING:
Plan to Share IPD: No